CLINICAL TRIAL: NCT05957835
Title: The Effect of Beetroot Juice Supplementation Dose on Neuromuscular Performance During Resistance Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pepperdine University (Other)
Responsible Party: Principal Investigator, Rachel Tan, Assistant Professor of Sports Medicine, Pepperdine University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: RT12
Record Dates: First submitted 2023-06-28; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: High Nitrate Dose; Moderate Nitrate Dose; Low Nitrate Dose; Nitrate-depleted Dose

STUDY DESIGN:
Intervention Model Description: In a double-blind, randomised, crossover design, participants were assigned to four experimental trials to consume a total of 4 beetroot juice shots during each condition: (a) 4 x 70 ml of nitrate-depleted beetroot juice for placebo (PL), (b) 1 x 70 ml of nitrate-rich beetroot juice 3 x 70 ml nitrate-depleted beetroot juice for a low dose of nitrate-rich beetroot juice (BR-LOW; ~6.5 mmol of nitrate total), (c) 2 x 70 of nitrate-rich beetroot juice and 2 x 70ml of nitrate depleted beetroot juice for a moderate dose of nitrate-rich beetroot juice (BR-MOD; ~13 mmol of nitrate total), and (d) 4 x 70 ml of nitrate-rich beetroot juice for an elevated dose of nitrate-rich beetroot juice (BR-HIGH; ~26 mmol of nitrate total).
Who Masked: Participant, Outcomes Assessor
Masking Description: The lead researcher, data collectors, and participants were blinded to the conditions. The distribution of supplements for each condition was performed by a researcher that was not formally involved in data collection processes, thereby limiting the potential of bias.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BR-HIGH (Experimental): Participants will ingest an elevated dose of nitrate 2.5 hours prior to exercise.
  Interventions: Dietary Supplement: BR-HIGH
- BR-MOD (Experimental): Participants will ingest a moderate dose of nitrate 2.5 hours prior to exercise.
  Interventions: Dietary Supplement: BR-MOD
- BR-LOW (Experimental): Participants will ingest a low dose of nitrate 2.5 hours prior to exercise.
  Interventions: Dietary Supplement: BR-LOW
- PL (Placebo Comparator): Participants will ingest a negligible amount of nitrate 2.5 hours prior to exercise.
  Interventions: Dietary Supplement: PL

INTERVENTIONS:
Dietary Supplement: BR-HIGH — 4 x nitrate-rich beetroot juice shots (26 mmol of nitrate)
  Arms: BR-HIGH
Dietary Supplement: BR-MOD — 2 x nitrate-rich beetroot juice shots + 2 x nitrate-depleted beetroot juice shot (12 mmol of nitrate)
  Arms: BR-MOD
Dietary Supplement: BR-LOW — 1 x nitrate-rich beetroot juice shot + 3 x nitrate-depleted beetroot juice shots (6 mmol of nitrate)
  Arms: BR-LOW
Dietary Supplement: PL — 4 x nitrate-depleted beetroot juice shots (0 mmol of nitrate)
  Arms: PL

SUMMARY:
Dietary nitrate supplementation, administered in the form of nitrate-rich beetroot juice, has been shown to improve exercise performance and may have more pronounced effects on exercise that requires high-power and high-velocity muscle contraction such as weightlifting and body-mass resisted exercise (i.e, resistance exercise). However, limited data are available that have examined the potential performance enhancing effect of beetroot juice in resistance exercise. Moreover, there is no information on the dose of nitrate required for performance enhancing effects during resistance exercise which limits its widespread use to enhance performance. Therefore, the investigators will assess if supplementing the diet with nitrate-rich beetroot juice impacts resistance exercise performance (e.g., power, velocity), when compared to supplementing the diet with nitrate-depleted beetroot juice (i.e. placebo). The investigators will also investigate the dose-response effect of beetroot juice on resistance exercise performance by providing a low, moderate, and high nitrate dose of concentrated beetroot juice. The results of this study will improve understanding of whether beetroot juice influences resistance exercise performance and will provide insight on whether different doses of beetroot juice influence the efficacy of nitrate supplementation on resistance exercise performance. Together, these data will guide supplementation strategies for enhancing resistance exercise performance.

DETAILED DESCRIPTION:
Supplementation with inorganic nitrate, which is most commonly administered in the form of concentrated nitrate-rich beetroot juice shots, has emerged as an ergogenic nutritional strategy. Beetroot juice ingestion has been reported to enhance endurance and high-intensity intermittent exercise performance in running and cycling. These improvements are attributed to augmented muscle contractility, force production and blood flow distribution, specifically in muscle groups comprised predominantly of type II muscle fibers. Together, such changes provide a strong physiological rationale supporting the potential for dietary nitrate to enhance high-power and high-velocity muscle contractions since type II muscle fibers are heavily activated during these tasks. However, the influence of dietary nitrate on resistance exercise performance is substantially underdeveloped with most previous studies having assessed the effect of nitrate supplementation on running and cycling endurance and high-intensity intermittent exercise. Moreover, there is no information on the dose of nitrate required to evoke ergogenic effects during resistance exercise, which greatly hinders the potential implementation of beetroot juice as a research-informed performance enhancing supplement for resistance exercise. Thus, the proposed project will investigate if acute dietary nitrate ingestion, provided as nitrate-rich beetroot juice, elicits improvements in various neuromuscular performance parameters (e.g., power, velocity) during resistance exercise performance when compared to supplementing the diet with a nitrate-depleted beetroot juice placebo. The investigators will also investigate the dose-response effect of beetroot juice on resistance exercise performance by providing low (70 ml i.e., ~6.5 mmol or ~400 mg of nitrate), moderate (140 ml i.e., ~13 mmol or ~800 mg of nitrate) and a high nitrate dose (280 ml i.e., ~26 mmol or ~1600 mg of nitrate) of concentrated beetroot juice. This project will provide insight to practitioners (coaches/athletes) aiming to enhance performance in settings where muscular power and speed are key determinants for success, as well as to scientists exploring the efficacy of beetroot juice as a form of dietary nitrate supplementation to improve muscle contractile function.

ELIGIBILITY:
Inclusion Criteria:

* Recreationally active males who performed resistance exercise at least twice weekly for the last two years

Exclusion Criteria:

* individuals with contraindications to exercise, cardiometabolic disease, currently consuming dietary supplements containing caffeine, sodium bicarbonate, creatine, beta-alanine, and/or NO precursor supplements (i.e., NO3-, arginine, citrulline, antioxidants), females, and smokers

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females were excluded given that sex-differences in the physiological responses to nitrate ingestion may exist and that including the appropriate controls (i.e., testing only during the early follicular phase) would have been unfeasible logistically.
Enrollment: 18 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-28 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Plasma nitrate | Through study completion, at least 1 year
  Plasma nitrate concentrations in each condition from blood samples draw at rest prior to exercise, and analyzed using gas phase chemiluminescence
Plasma nitrite | Through study completion, at least 1 year
  Plasma nitrite concentrations in each condition from blood samples draw at rest prior to exercise, and analyzed using gas phase chemiluminescence
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  Peak force will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  average propulsion force will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  rate of power development will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  peak positive power will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  concentric mean power will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  jump height will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  takeoff velocity will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  flight time will be measured using a force place.
Neuromuscular performance during countermovement jumps | Through study completion, at least 1 year
  Peak force, average propulsion force, rate of power development, peak positive power, concentric mean power, jump height, takeoff velocity, flight time will be measured using a force place.
Peak power | Through study completion, at least 1 year
  Power will be measured using a linear transducer with the highest value will be recorded for peak power
Mean power | Through study completion, at least 1 year
  Power will be measured using a linear transducer and will be averaged across sets for the determination of mean power
Mean velocity | Through study completion, at least 1 year
  Velocity will be measured using a linear transducer and will be averaged across sets for the determination of mean velocity
Peak velocity | Through study completion, at least 1 year
  Velocity will be measured using a linear transducer the highest value will be retained for peak velocity

SECONDARY OUTCOMES:
Mood | Through study completion, at least 1 year
  24 items representing six subscales (i.e., anger, confusion, depression, fatigue, tension, vigour; four-items per subscale) will be captured using a five-point Likert scale (i.e., 0 = not at all, 1 = a little, 2 = moderately, 3 = quite a bit, 4 = extremely)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Tan, PhD, Principal Investigator — Pepperdine University
Locations (1):
- Pepperdine University, Malibu, California, United States

IPD SHARING:
Plan to Share IPD: No
The raw data supporting the conclusions of this article will be made available by the authors, without undue reservation, upon request.